CLINICAL TRIAL: NCT01591434
Title: An Open Randomised Comparative Study to Evaluate the Performance of AQUACEL® Extra™ in Venous Leg Ulcers
Brief Title: Study to Evaluate the Performance of AQUACEL® Extra™ in Venous Leg Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CW-0209-11-U361
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Leg Ulcer
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AQUACEL® (Active Comparator): A sterile non-woven sheet of sodium carboxymethylcellulose (NaCMC).
  Interventions: Device: AQUACEL®
- AQUACEL® Extra™ (Active Comparator): A sandwiched construction of two layers of optimally textiled non-woven fabric, stitch-bonded together using Lyocel (Tencel™ regenerated cellulose) yarns.
  Interventions: Device: AQUACEL® Extra™

INTERVENTIONS:
Device: AQUACEL® — Dressing to be changed as clinically needed or at least every seven days.
  Arms: AQUACEL®
Device: AQUACEL® Extra™ — Dressing to be changed as clinically needed or at least every seven days.
  Arms: AQUACEL® Extra™

SUMMARY:
Based upon the in-vitro data AQUACEL® Extra™ achieves a 39% increase in absorbency. As such it is anticipated that through improved exudate management a longer wear time will be achieved in the AQUACEL® Extra™ group compared to AQUACEL® in the management of chronic wounds such as venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years, willing and able to provide written informed consent.
* Subjects who have an ankle to brachial pressure index (ABPI) of 0.8 or greater
* Subjects who have a venous leg ulcer (i.e. CEAP classification of C6 1) with duration less than 24 months
* Subjects whose ulcer is no smaller than 2cms in any one direction
* Subjects whose ulcer is no greater than 11cm in any one direction (measured by longest length and widest width)
* Subjects' whose index leg ulcer has a moderate to heavy level of exudate.
* Subjects whose index (study) leg is currently being treated with compression therapy and whose leg oedema is under control
* Subjects who are willing and able to comply with the requirements of the clinical investigation plan in relation to the dressing/compression regime and the ability to attend dressing changes as required.

Exclusion Criteria:

* Subjects with a history of skin sensitivity to any of the components of the study dressings (AQUACEL® Extra™, AQUACEL®, & DuoDERM™ Extra Thin)
* Subjects whose wounds are considered clinically infected at baseline
* Subjects whose leg ulcers are malignant, or who have had recent deep venous thrombosis or venous surgery within the last 3 months.
* Subjects who have progressive neoplastic lesion treated by radiotherapy or chemotherapy, or on-going treatment with immunosuppressive agents
* Subjects exhibiting any other medical condition which, according to the Investigator, justifies the subject's exclusion from the study
* Subjects who have participated in a clinical study within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Wear Time | 4 weeks
  frequency of dressing changes
Wear Time | 4 weeks
  Reason for dressing changes
% of dressings achieving a 7 day wear time | 4 weeks
Time to achieve a 7 day wear time | 4 weeks
Condition of the peri-ulcer skin | 4 weeks
  Improvement from baseline in the condition of the peri-ulcer skin

CONTACTS AND LOCATIONS:
Overall Officials: Keith G Harding, Principal Investigator — Cardiff University
Locations (12):
- Germany (2):
  - Dermatologische Gemeinschaftspraxis, Freiburg im Breisgau
  - Bramfelder Chaussee, Hamburg
- Mitralis Expertise Centrum, Heerlen, Netherlands
- Poland (4):
  - Nzoz Certus, Lodz
  - CF Centrum Flebologii Anna i Beata Narojczyk, Warsaw
  - Continuum Care, Warsaw
  - Medyczna "Medservice", Zabrze
- United Kingdom (5):
  - Arrowe Park Hospital,, Upton, Wirral
  - Bradford Teaching Hospitals, Bradford
  - Wound Healing Research Unit, Cardiff University, Cardiff
  - Tissue Viability Consultancy Services Ltd, Eastbourne
  - Walsall Healthcare NHS Trust Short Heath Clinic, Willenhall